CLINICAL TRIAL: NCT06595420
Title: Kidney Function in People With Cystic Fibrosis in the Era of HEMT
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Agnieszka Swiatecka-Urban, Professor of Pediatrics, University of Virginia
Other Study IDs: HSR231650; 005245A123 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis (CF); Chronic Kidney Disease(CKD); Acute Kidney Injury
MeSH Terms: conditions — Cystic Fibrosis; Renal Insufficiency, Chronic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Outpatient CF Cohort: Not hospitalized CF group: Diagnosis of CF, age >30 y, with ongoing care at one of the 3 CF Centers (Dartmouth, UAB, UVA).
- Inpatient CF Cohort: Hospitalized CF cohort: Diagnosis of CF, age >7 y, being admitted for intravenous antibiotic treatment of pulmonary exacerbation.
- Healthy Controls: Healthy Volunteers without CF

SUMMARY:
The purpose of this study is to find out what causes kidney disease in people with CF. The investigators will study biomarkers in the blood and urine that can either predict who is at risk or detect kidney damage early before it becomes permanent. The study will compare these markers in people with CF over time and during the treatment of lung flare-ups. It will also compare the blood and urine samples obtained from people without CF. The comparison aims to better understand the impact of cystic fibrosis and its treatment on the kidneys, as well as to develop improved methods for preventing, diagnosing, and treating kidney issues associated with CF.

DETAILED DESCRIPTION:
The prevalence of chronic kidney disease is significantly increased in patients with cystic fibrosis (PwCF) with a major impact on morbidity and medication tolerance as people age. Although expressed in both the proximal and distal tubules, the specific contribution of CFTR dysfunction to renal disease remains uncertain. PwCF often are exposed to renal toxins such as frequent aminoglycosides, systemic inflammation, and activated leukocytes, but it is unknown if CFTR dysfunction predisposes to amplified tubular injury. Conventional measures of kidney function, such as serum creatinine, are insensitive to detecting early injury, limiting an opportunity to prevent CKD. This study will address the gaps in early detection and mechanisms of renal dysfunction in CF. The investigators will define the triggers and targetable mechanistic pathways of kidney injury in CF and discover novel strategies for renal protection. The central hypothesis of this study is that CFTR dysfunction alters renal development and increases the inflammatory and fibrogenic responses to nephrotoxic stimuli.

The study involves prospective evaluation of biospecimens (blood and urine) and clinical data. The study analyzes biospecimens in CF outpatients (n=110), CF inpatients (n=110), and healthy subjects (n=40). In the outpatient cohort, biospecimens will be collected at the time of each routine care visit every 3 months for 24 months. PwCF admitted for intravenous (IV) antibiotics will have biospecimens collected on admission and every 48 hrs thereafter during the admission, and then after hospital discharge at each subsequent clinical encounter for 24 months.

These biospecimens will be analyzed for biomarkers, fibrogenic analysis, inflammatory signals, and extracellular vesicles. Clinical data will be examined from chart review and correlated with biospecimen result.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient CF Cohort

   * Diagnoses of Cystic Fibrosis
   * Age > 30 years old
   * Able to provide informed consent
2. Inpatient CF Cohort

   * Diagnoses of Cystic Fibrosis
   * Age > 7 years old
   * Able to provide informed consent and assent (where applicable)
   * 55 PwCF frequently hospitalized for a pulmonary exacerbation (>1 hospital admission in the prior 12 months)
   * 55 PwCF sporadically hospitalized for a pulmonary exacerbation (no hospital admissions in the prior 12 months)
   * Able to provide urine sample independently
3. Healthy Controls

   * Healthy, as per participant self-report
   * Age between 30-50 years
   * Able to provide informed consent

Exclusion Criteria:

1. Outpatient CF Cohort

   * History of any organ transplant
   * History of immunodeficiency
   * Previous or current cancer diagnoses
   * Pregnant or breastfeeding
   * On chronic dialysis
   * Non-compliance (demonstrated by <2 visits during the 12 months before enrollment)
2. Inpatient CF Cohort

   * The initiation of intravenous antibiotic therapy after hospital admission before obtaining the first blood and urine sample
   * History of any organ transplant
   * History of immunodeficiency
   * Previous or current cancer diagnoses
   * Pregnant or breastfeeding
   * On chronic dialysis
3. Healthy Controls

   * History or current kidney disease, organ transplantation, cancer, or any other chronic illness
   * Current use of antibiotics
   * Urinary symptoms or UTI (dysuria, frequency, urgency)
   * Pregnant women
   * Menstruating on the study visit day
   * Blood relatives of PwCF

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be derived from patients with CF with ongoing care at one of the 3 CF Centers (Dartmouth, UAB, UVA).
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Examine whether trajectories of eGFR (calculated from serum creatinine and cystatin C) correlate with urinary kidney injury signatures detected in different urine fractions, or urinary neutrophil levels/activation. | Enrollment and every 3 months for 24 months
  Outpatient CF Cohort
Correlation between recurrent hospitalizations and urinary kidney injury signature. | On admission before the initiation of intravenous antibiotic therapy, every 48 hrs during the hospitalization, after discharge at each subsequent routine CF care visit for 24 months.
  Inpatient CF Cohort
Relationship between recurrent hospitalization and change in slope of eGFR | On admission before the initiation of intravenous antibiotic therapy, every 48 hrs during the hospitalization, after discharge at each subsequent routine CF care visit for 24 months.
  Inpatient CF Cohort

SECONDARY OUTCOMES:
The correlation between changes in the urinary protein biomarker panel, neutrophil activation, and extracellular vesicles over time and eGFR. | Enrollment and every 3 months for 24 months.
  Outpatient CF Cohort
Correlation between %FEV1 at admission or decline in %FEV1 and urinary kidney injury signature. | On admission before the initiation of intravenous antibiotic therapy, every 48 hrs during the hospitalization, after discharge at each subsequent routine CF care visit for 24 months.
  Inpatient CF Cohort

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Dartmouth-Hitchcock Geisel School of Medicine at Dartmouth, Lebanon, New Hampshire
  - University of Virginia Children's Hospital, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devuyst O, Burrow CR, Schwiebert EM, Guggino WB, Wilson PD. Developmental regulation of CFTR expression during human nephrogenesis. Am J Physiol. 1996 Sep;271(3 Pt 2):F723-35. doi: 10.1152/ajprenal.1996.271.3.F723. PMID 8853436
- [Background] Southern KW. Acute renal failure in people with cystic fibrosis. Thorax. 2007 Jun;62(6):472-3. doi: 10.1136/thx.2006.072355. PMID 17536029
- [Background] Al-Aloul M, Miller H, Alapati S, Stockton PA, Ledson MJ, Walshaw MJ. Renal impairment in cystic fibrosis patients due to repeated intravenous aminoglycoside use. Pediatr Pulmonol. 2005 Jan;39(1):15-20. doi: 10.1002/ppul.20138. PMID 15521084
- [Background] Bertenshaw C, Watson AR, Lewis S, Smyth A. Survey of acute renal failure in patients with cystic fibrosis in the UK. Thorax. 2007 Jun;62(6):541-5. doi: 10.1136/thx.2006.067595. Epub 2007 Jan 18. PMID 17234661
- [Background] Quon BS, Mayer-Hamblett N, Aitken ML, Smyth AR, Goss CH. Risk factors for chronic kidney disease in adults with cystic fibrosis. Am J Respir Crit Care Med. 2011 Nov 15;184(10):1147-52. doi: 10.1164/rccm.201105-0932OC. Epub 2011 Jul 28. PMID 21799076
- [Background] Stevanovic M, G.M. Primary Causes of ESRD in the US Cystic Fibrosis Population. JASN 33, 694
- [Background] Stevanovic, M.G.M.L. Characteristics of US Individuals with Cystic Fibrosis and ESRD. JASN 33, 694
- [Background] Lai S, Mazzaferro S, Mitterhofer AP, Bonci E, Marotta PG, Pelligra F, Murciano M, Celani C, Troiani P, Cimino G, Palange P. Renal involvement and metabolic alterations in adults patients affected by cystic fibrosis. J Transl Med. 2019 Nov 25;17(1):388. doi: 10.1186/s12967-019-02139-4. PMID 31767021
- [Background] Berg KH, Ryom L, Faurholt-Jepsen D, Pressler T, Katzenstein TL. Prevalence and characteristics of chronic kidney disease among Danish adults with cystic fibrosis. J Cyst Fibros. 2018 Jul;17(4):478-483. doi: 10.1016/j.jcf.2017.11.001. Epub 2017 Dec 1. PMID 29187303
- [Background] Alicandro G, Frova L, Di Fraia G, Colombo C. Cystic fibrosis mortality trend in Italy from 1970 to 2011. J Cyst Fibros. 2015 Mar;14(2):267-74. doi: 10.1016/j.jcf.2014.07.010. Epub 2014 Aug 20. PMID 25151032
- [Background] Nazareth D, Walshaw M. A review of renal disease in cystic fibrosis. J Cyst Fibros. 2013 Jul;12(4):309-17. doi: 10.1016/j.jcf.2013.03.005. Epub 2013 Apr 22. PMID 23618617
- [Background] van Duijl TT, Ruhaak LR, de Fijter JW, Cobbaert CM. Kidney Injury Biomarkers in an Academic Hospital Setting: Where Are We Now? Clin Biochem Rev. 2019 May;40(2):79-97. doi: 10.33176/AACB-18-00017. PMID 31205376
- [Background] Kovesdy CP, Bleyer AJ, Molnar MZ, Ma JZ, Sim JJ, Cushman WC, Quarles LD, Kalantar-Zadeh K. Blood pressure and mortality in U.S. veterans with chronic kidney disease: a cohort study. Ann Intern Med. 2013 Aug 20;159(4):233-42. doi: 10.7326/0003-4819-159-4-201308200-00004. PMID 24026256
- [Background] Breyer MD, Susztak K. The next generation of therapeutics for chronic kidney disease. Nat Rev Drug Discov. 2016 Aug;15(8):568-88. doi: 10.1038/nrd.2016.67. Epub 2016 May 27. PMID 27230798
- [Background] Kovesdy CP. Epidemiology of chronic kidney disease: an update 2022. Kidney Int Suppl (2011). 2022 Apr;12(1):7-11. doi: 10.1016/j.kisu.2021.11.003. Epub 2022 Mar 18. PMID 35529086